CLINICAL TRIAL: NCT05814744
Title: Efficacy of Adding Dexmedetomidine as Adjuvant With Bupivacaine in Ultrasound-guided Intermediate Cervical Plexus Block for Thyroidectomy Surgery: Randomized Controlled Study
Brief Title: Efficacy of Adding Dexmedetomidine in Ultrasound-guided Intermediate Cervical Plexus Block for Thyroidectomy Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Cancer Institute, Egypt (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: AP2211-301-045
Record Dates: First submitted 2023-02-21; First posted 2023-04-18 (Actual); Last update posted 2024-04-05 (Actual); Status verified 2023-04

CONDITIONS: Pain, Postoperative; Cancer of Larynx
Keywords: Intermediate Cervical Plexus Block; dexmedetomidine; bupivacaine; Thyroidectomy surgery
MeSH Terms: conditions — Pain, Postoperative; Laryngeal Neoplasms | interventions — Dexmedetomidine; Bupivacaine

STUDY DESIGN:
Intervention Model Description: randomized
Who Masked: Participant, Investigator
Masking Description: double blind
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group (A) (Sham Comparator): bupivacaine 0.25% only
  Interventions: Drug: bupivacaine 0.25%; Procedure: Thyroidectomy Surgery; Procedure: Ultrasound-guided intermediate Cervical Plexus Block Technique
- Group (B) (Active Comparator): bupivacaine 0.25% and dexmedetomidine
  Interventions: Drug: dexmedetomidine; Drug: bupivacaine 0.25%; Procedure: Thyroidectomy Surgery; Procedure: Ultrasound-guided intermediate Cervical Plexus Block Technique

INTERVENTIONS:
Drug: dexmedetomidine — adding dexmedetomidine as adjuvant with bupivacaine in Ultrasound-guided Intermediate Cervical Plexus Block for Thyroidectomy surgery.
  Other Names: precedex vial
  Arms: Group (B)
Drug: bupivacaine 0.25% — patients will receive bilateral Intermediate Cervical plexus block with 20 ml bupivacaine 0.25%.
  Other Names: Sensorcaine®
Procedure: Thyroidectomy Surgery — surgical removal of all or part of thyroid gland.
Procedure: Ultrasound-guided intermediate Cervical Plexus Block Technique — the injection of local anesthetic in intermediate cervical plexus nerve block is made between the investing layer of the deep cervical fascia and the prevertebral fascia. Following negative aspiration, 1-2 mL of local anesthetic is injected to confirm the proper injection site.

SUMMARY:
The cervical plexus block (CPB) is one such block used to provide effective anesthesia and analgesia for surgery in the head and neck region. The cervical fascia was first described as a very strong and resisting structure, consisting of two layers, superficial and deep. But more recently classified the cervical fascia as superficial/subcutaneous and deep. The deep cervical fascia is further divided into three layers: (a) the superficial layer, which was also called the investing fascia but is now referred to as the masticator fascia, submandibular fascia or sternocleidomastoid (SCM)-trapezius fascia, (b) the middle layer, which is suggested as to be named as strap muscle fascia or visceral fascia; and (c) the deep layer or the 'prevertebral fascia'. Intermediate cervical plexus block (CPB) has been found to be very effective in procedures of neck such as thyroid surgeries and carotid endarterectomy. The duration of analgesia following the nerve blocks is a matter of concern as most of the blocks last for only a few hours. Interestingly, resurgence of the use of α2-agonists in combination with local anesthetics has dramatically improved the duration of action of these blocks. Dexmedetomidine is a potent α2 agonist and is now emerging as an adjuvant to regional anesthesia and analgesia. Little evidence is available supporting the usefulness of dexmedetomidine in bilateral intermediate CPB. Therefore, the current study will be conducted to compare the duration and effectiveness of post-thyroidectomy analgesia of bilateral intermediate CPB using 20 ml bupivacaine 0.25% (Group A) or 20 ml of bupivacaine 0.25% with 1 μg/kg dexmedetomidine (Group B).

DETAILED DESCRIPTION:
- Objectives: The aim of this study is to evaluate the effect of adding dexmedetomidine as adjuvant to bupivacaine in ultrasound guided Intermediate Cervical Plexus Block (CPB) for thyroidectomy surgery.

- Study Design : Double-blind randomized controlled study where both patient and investigator don't know the drug.

- Study Methodology:

1. Population of study & disease Condition Adult patients at National Cancer Institute scheduled for thyroidectomy fulfilling the eligibility criteria.
2. Interventions:

   All patients will be medically checked in the preoperative assessment clinic {history, physical examination, investigations (e.g., complete blood picture, coagulation profile, liver & kidney functions, ECG for patients above 40 years, pulmonary function test (PFT) and any other necessary investigations if required for high-risk patients.)} Preoperative assessment at night of surgery. The patients will be instructed how to report pain by means of visual analogue scale [VAS] during the preoperative assessment. Informed consent will be obtained.

   In the holding room, the patients will be continuously monitored for pulse, blood pressure, oxygen saturation. Intravenous (IV) 18-gauge cannula will be inserted for all patients. Midazolam 0.02 mg/Kg will be administered. For each patient, 7-10 ml/kg of intravenous (IV) ringer acetate will be administered if required to replace fluid deficiency 30 min before the surgery. Portable ultrasound machine, resuscitation equipment &drugs (e.g., epinephrine, lipid emulsion), sterile gloves and surgical towels should be available.

   Anesthetic Management:

   Monitoring: all patients will be monitored continuously using ECG, Non Invasive Blood Pressure (NIBP), peripheral arterial oxygen saturation and end tidal carbon dioxide throughout the duration of surgery. Regimen of IV 2 μg/kg fentanyl and propofol IV 2 mg /kg will be used for Induction of general anesthesia. Tracheal intubation will be facilitated using 0.5 mg/kg IV of rocuronium. After Induction of general anesthesia (GA) both groups' patients will receive bilateral Intermediate Cervical plexus block, either with 20 ml bupivacaine 0.25% (Group A) or 20 ml of bupivacaine 0.25% with 1 μg/kg dexmedetomidine (Group B). Anesthesia will be maintained with inhaled sevoflurane with minimum alveolar concentration (MAC) 2-2.5% in oxygen enriched air (FiO2=50%) and top up doses of rocuronium (0.1 mg/kg) IV will be administered as required. All patients will receive 1 g of IV paracetamol.

   Additional bolus doses of fentanyl 0.5 µg/kg will be given if the mean arterial blood pressure or heart rate rises above 20% of baseline levels.

   At the end of surgery, the residual neuromuscular blockade will be reversed using neostigmine (0.05 mg/kg) and atropine (0.02 mg/kg), and extubation will be performed after complete recovery of the airway reflexes.

   After surgery the patients will be transferred to the post anesthesia care unit where pain scores and mean arterial pressure (MAP) and heart rate will be noted immediately on arrival and at 2, 4, 6, 12 and 24 hours postoperatively. The patients will be observed in the postoperative care unit for 2 h, and rescue analgesia will be provided in the form of IV morphine 3 mg boluses if the pain score >3. The total amount of morphine given in 24 hours will be recorded in the two groups. Thereafter, the patients will be shifted to ward and will be given acetaminophen 1 g IV every 8 hours.

   Ultrasound-guided intermediate cervical plexus block (CPB) Technique:

   The block is performed with full aseptic precautions. The block is performed in the supine position, the head is turned to the opposite side and. The patient's neck and upper chest should be exposed so that the relative length and position of the SCM can be assessed.

   The skin is disinfected and the transducer is placed on the lateral neck, overlying the SCM at the level of its midpoint (approximately the level of the cricoid cartilage).

   Once the SCM has been identified, the transducer is moved posteriorly until the tapering posterior edge is positioned in the middle of the screen. At this point, an attempt should be made to identify the brachial plexus and/or the interscalene groove between the anterior and middle scalene muscles. The cervical plexus is visible as a small collection of hypoechoic nodules (honeycomb appearance) immediately superficial to the prevertebral fascia that overlies the interscalene groove.

   Once the plexus has been identified, local anesthetic (LA) can be injected using long axis, in plane approach by keeping the probe in transverse position. For intermediate cervical plexus nerve block, the injection is made between the investing layer of the deep cervical fascia and the prevertebral fascia. Following negative aspiration, 1-2 mL of local anesthetic is injected to confirm the proper injection site. The remainder of the local anesthetic is administered to envelop the plexus.
3. Possible Risk and Adverse events:

   1. Failure of block.
   2. Local anesthetic toxicity.

f) Sample size (number of participants included approved by statistical calculation

A recent randomized double blinded study showed that US-guided intermediate cervical plexus block (CPB) was better than superficial CBP for post-operative analgesia in patients undergoing total thyroidectomy. On the other-hand a randomized double blinded study found that adding dexmedetomidine to superficial CPB improve analgesia for thyroid surgeries. Based on the results (evidences) of previous study on the evidence that intermediate CPB is better than superficial CBP for post-operative analgesia the investigators based the calculation of sample size for the current study.

In this study, they found that for the patients' group where CPB is done with 20 ml 0.5% ropivacaine (Group A) or 20 ml 0.5% ropivacaine with 0.5 µg/kg dexmedetomidine (Group B) the following was found:

1. Longer duration of analgesia in group B than group A (1696.2±100.2 minutes and 976.8±81.6 minutes respectively, p <0.001).
2. Median VAS score at 12 hours postoperatively was 2(1-2) in group A vs 0(0-1) in group B, and median VAS score at 24 hours postoperatively was 5(5-6) in group A vs 2(2-2) in group B, p < 0.001.

Based on the above estimates for duration of analgesia and VAS scores in both groups, sample size was calculated with these expected means (or medians as an approximate estimate) and a pooled standard deviation SD (being always conservative and taking the largest SD), assuming a power of 95% and level of significance of 0.01, maximum sample size needed per group was 5 with a total of 10 patients to find the above differences between the two groups with the power and significance described. As the investigators want to assume normality of variables as VAS score, sample size was corrected to be 30 per group with a total of 60 patients to be equally and randomly allocated to either group receiving bupivacaine alone or with dexmedetomidine.

Randomization was done using SPSS , table of random allocation of the two study groups.

d) Statistical analysis of data:

Data will be collected from patients and tabulated using SPSS version 23.0 (SPSS inc., Chicago, USA). Quantitative data will be presented as mean and standard deviation if found normally distributed and median and range if else. Parametric and non-parametric t-test will compare means of two independent groups such as age, weight, duration of analgesia, vitals of the patients, VAS score …etc. Rates of complications will be compared using Chi-square or Fisher exact tests. P value will be considered significant if ≤0.05 and will be always two tailed.

e) Source of funding:

Funded by National Cancer Institute, Cairo University.

ELIGIBILITY:
Inclusion Criteria:

* Physical status American society Anesthesiologists ASA II and III.
* Age ≥ 18 and ≤ 60 Years.
* Patient undergoing thyroidectomy for cancer surgery.

Exclusion Criteria:

* Patient refusal.
* Known sensitivity or contraindication to local anesthetics or dexmedetomidine.
* History of psychological disorders.
* Retro-sternal goiter and altered anatomical landmarks.
* Localized infection at the site of block.
* Coagulopathy with international normalized ratio (INR) ≥ 1.6: hereditary (e.g., hemophilia, fibrinogen abnormalities & deficiency of factor II) - acquired (e.g., impaired liver functions with prothrombin concentration less than 60 %, vitamin K deficiency & therapeutic anticoagulants drugs).

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2023-04-01 (Actual); Primary Completion 2023-10-01 (Actual); Study Completion 2023-11-01 (Actual)

PRIMARY OUTCOMES:
first rescue analgesia | the first 24 hours of postoperative period
  First time (minutes) opioids requested postoperative when pain score is >3 .

SECONDARY OUTCOMES:
Total intraoperative fentanyl consumption. | throughout the duration of the surgery
  the doses of fentanyl will be given if the mean arterial blood pressure or heart rate rises above 20% of baseline levels.
postoperative opioids consumption. | 24 hours postoperative
  Total patient's morphine requirements within 24 hours postoperative.
Post-operative pain scores. | immediately postoperative (0 hours ), 2, 4, 6, 12 and 24 hours postoperative
  Post-operative pain scores using Visual analogue score (VAS) (0 mm = no pain to 10mm = worst pain imaginable) at predetermined time intervals
Any complications will be recorded. | throughout the duration of the surgery and 24 hours postoperative
  Any complications such as failed block, hypotension, unintentional intravascular injection of LA and local anesthetic toxicity will be recorded.

CONTACTS AND LOCATIONS:
Overall Officials: Gehan M. Kamal, Prof., Principal Investigator — National Cancer Institute, Anesthesia, Pain Relief and ICU Department; Mohamed E. Hassan, Ass. Prof., Principal Investigator — National Cancer Institute, Anesthesia, Pain Relief and ICU Department; Mai M. Elrawas, Doctor, Principal Investigator — National Cancer Institute, Anesthesia, Pain Relief and ICU Department
Locations (1):
- National Cancer Institue, Cairo, Fom El Khalig, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Syal K, Chandel A, Goyal A, Sharma A. Comparison of ultrasound-guided intermediate vs subcutaneous cervical plexus block for postoperative analgesia in patients undergoing total thyroidectomy: A randomised double-blind trial. Indian J Anaesth. 2020 Jan;64(1):37-42. doi: 10.4103/ija.IJA_483_19. Epub 2020 Jan 7. PMID 32001907
- [Background] Natale G, Condino S, Stecco A, Soldani P, Belmonte MM, Gesi M. Is the cervical fascia an anatomical proteus? Surg Radiol Anat. 2015 Nov;37(9):1119-27. doi: 10.1007/s00276-015-1480-1. Epub 2015 May 7. PMID 25946970
- [Background] Guidera AK, Dawes PJ, Fong A, Stringer MD. Head and neck fascia and compartments: no space for spaces. Head Neck. 2014 Jul;36(7):1058-68. doi: 10.1002/hed.23442. Epub 2014 Jan 29. PMID 23913739
- [Background] Kim, J.-S. and H.Y. Kim, Cervical plexus block. Surgical Anatomy of the Cervical Plexus and its Branches, 2022: p. 189-202.
- [Background] Egan RJ, Hopkins JC, Beamish AJ, Shah R, Edwards AG, Morgan JD. Randomized clinical trial of intraoperative superficial cervical plexus block versus incisional local anaesthesia in thyroid and parathyroid surgery. Br J Surg. 2013 Dec;100(13):1732-8. doi: 10.1002/bjs.9292. PMID 24227357
- [Background] Kaygusuz K, Kol IO, Duger C, Gursoy S, Ozturk H, Kayacan U, Aydin R, Mimaroglu C. Effects of adding dexmedetomidine to levobupivacaine in axillary brachial plexus block. Curr Ther Res Clin Exp. 2012 Jun;73(3):103-11. doi: 10.1016/j.curtheres.2012.03.001. PMID 24648597
- [Background] Andersen JH, Grevstad U, Siegel H, Dahl JB, Mathiesen O, Jaeger P. Does Dexmedetomidine Have a Perineural Mechanism of Action When Used as an Adjuvant to Ropivacaine?: A Paired, Blinded, Randomized Trial in Healthy Volunteers. Anesthesiology. 2017 Jan;126(1):66-73. doi: 10.1097/ALN.0000000000001429. PMID 27792047
- Available data/document: Individual Participant Data Set — https://drive.google.com/file/d/12gNVWYJj8dyy6Bh-6G59rFn2AQzjHycS/view?usp=share_link
- Available data/document: Informed Consent Form — https://drive.google.com/file/d/1qPpYheG63CcWJqwWAD3ma3jFmmqCPWgm/view?usp=share_link
- Available data/document: Study Protocol — https://drive.google.com/file/d/16x_dHL6GsO6V-K3p13T9EluZi20l4WtN/view?usp=share_link